CLINICAL TRIAL: NCT01358097
Title: Biomarkers of Immune Function as Predictors of Head and Neck Squamous Cell Carcinoma (HNSCC) in Response to Therapy
Brief Title: Role of Immune Activation in Response of Head and Neck Squamous Cell Carcinoma to Therapy
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 10-1219
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Head and Neck Cancer; Oropharyngeal Cancer; Human Papillomavirus; Squamous Cell Cancer
Keywords: Head and neck cancer; Oropharyngeal cancer; Human papillomavirus; Squamous cell carcinoma; Radiation treatment; Chemotherapy; Induction chemotherapy; Immune status; Immune monitoring; head and neck robotic surgery
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms; Neoplasms, Squamous Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with HPV positive tumors
- Patients with HPV negative tumors
- Control

SUMMARY:
The purpose of this study is to investigate the role of the immune system in the response of squamous cell cancers of the head and neck to treatment that includes radiation therapy. Current research demonstrates that several natural immune cells and molecules affect the way the body's immune system interacts with a cancerous growth. Some cancers may be related to infection with a virus, such as the Human Papilloma Virus (HPV). Studying the activity of the immune system in head and neck cancers, especially cancers related to HPV infections, can provide valuable information to better understand the body's interaction with cancer cells.

DETAILED DESCRIPTION:
This is a study of the immune response in patients with oropharyngeal cancer who undergo treatment with radiation, chemoradiation, or robotic surgery. Many oropharyngeal cancers are caused by infection with the human Papillomavirus (HPV), and patients with HPV-mediated tumors have much better prognosis and treatment response compared to patients with HPV-negative tumors. The investigators will test the hypothesis that radiation-based therapy of oropharyngeal cancer is associated with activation of the endogenous HPV-specific immune response. In this study the investigators will collect blood at several time points before, during, and after treatment to monitor the immune response in patients with tumors positive and negative for HPV versus normal healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* The patient has biopsy-proven squamous cell carcinoma, Stage II-IV, of the oropharynx or larynx.
* The patient is to undergo treatment with radiation, chemo-radiation, or robotic surgery.
* The patient is able to give informed consent.
* The patient is at least 18 years old.
* The patient's ECOG performance status is </=2.

Exclusion Criteria:

* The patient has had prior head and neck squamous cell carcinoma, with the exception of superficial cutaneous basal cell or squamous cell carcinomas.
* The patient has active cancer in another part of the body, with the exception of superficial cutaneous basal cell or squamous cell carcinomas.
* If a cancer survivor, the disease free interval is less than 5 years, with the exception of superficial cutaneous basal cell or squamous cell carcinomas.
* The patient is a minor.
* The patient is pregnant.
* The patient is a prisoner.
* The patient is incapable of understanding the consent process.
* The patient has previously received definitive surgical, radiation, or chemoradiation treatment for HNSCC.
* The patient has a history of HIV or other known cause of immunosuppression, or is actively taking immunosuppressive medications due to organ transplantation, rheumatoid disease, or other medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with new head and neck cancer, who reside in the tri-state area.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2010-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
HPV-specific T-cell response | at time of enrollment into study (baseline)
HPV-specific T-cell response | after 3 weeks of treatment
HPV-specific T-cell response for HPV+ tumors | 3 months after completion of treatment
HPV-specific T-cell response for HPV+ tumors | 6 months after completion of treatment
HPV-specific T-cell response | 1 year after completion of treatment
HPV-specific T-cell response | 2 years after completion of treatment
HPV-specific T-cell response | 3 years after completion of treatment

SECONDARY OUTCOMES:
Circulating immune cells and cytokines | at time of enrollment into study (baseline)
Circulating immune cells and cytokines | after 3 weeks of treatment
Circulating immune cells and cytokines | 3 months after completion of treatment
Circulating immune cells and cytokines | 6 months after completion of treatment
Circulating immune cells and cytokines | one year after completion of treatment
Clinical outcome correlation | three years after treatment
inflammatory/regulatory cytokines | at time of enrollment (baseline)
inflammatory/regulatory cytokines | after 3 weeks of treatment
inflammatory/regulatory cytokines | 3 months after completion of treatment
inflammatory/regulatory cytokines | 6 months after completion of treatment
inflammatory/regulatory cytokines | 1 year after completion of treatment
serum nitrite/nitrate | after 3 weeks of treatment
serum nitrite/nitrate | 3 months after completion of treatment
serum nitrite/nitrate | 6 months after completion of treatment
serum nitrite/nitrate | 1 year after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sikora, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, Otolaryngology - Head and Neck Surgery, New York, New York, United States

REFERENCES:
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Estimating the world cancer burden: Globocan 2000. Int J Cancer. 2001 Oct 15;94(2):153-6. doi: 10.1002/ijc.1440. No abstract available. PMID 11668491
- [Background] Viale PH. The American Cancer Society's Facts & Figures: 2020 Edition. J Adv Pract Oncol. 2020 Mar;11(2):135-136. doi: 10.6004/jadpro.2020.11.2.1. Epub 2020 Mar 1. No abstract available. PMID 33532112
- [Background] Nasman A, Attner P, Hammarstedt L, Du J, Eriksson M, Giraud G, Ahrlund-Richter S, Marklund L, Romanitan M, Lindquist D, Ramqvist T, Lindholm J, Sparen P, Ye W, Dahlstrand H, Munck-Wikland E, Dalianis T. Incidence of human papillomavirus (HPV) positive tonsillar carcinoma in Stockholm, Sweden: an epidemic of viral-induced carcinoma? Int J Cancer. 2009 Jul 15;125(2):362-6. doi: 10.1002/ijc.24339. PMID 19330833
- [Background] Ringstrom E, Peters E, Hasegawa M, Posner M, Liu M, Kelsey KT. Human papillomavirus type 16 and squamous cell carcinoma of the head and neck. Clin Cancer Res. 2002 Oct;8(10):3187-92. PMID 12374687
- [Background] Fakhry C, Gillison ML. Clinical implications of human papillomavirus in head and neck cancers. J Clin Oncol. 2006 Jun 10;24(17):2606-11. doi: 10.1200/JCO.2006.06.1291. PMID 16763272
- [Background] Fakhry C, Westra WH, Li S, Cmelak A, Ridge JA, Pinto H, Forastiere A, Gillison ML. Improved survival of patients with human papillomavirus-positive head and neck squamous cell carcinoma in a prospective clinical trial. J Natl Cancer Inst. 2008 Feb 20;100(4):261-9. doi: 10.1093/jnci/djn011. Epub 2008 Feb 12. PMID 18270337
- [Background] Ang KK, Harris J, Wheeler R, Weber R, Rosenthal DI, Nguyen-Tan PF, Westra WH, Chung CH, Jordan RC, Lu C, Kim H, Axelrod R, Silverman CC, Redmond KP, Gillison ML. Human papillomavirus and survival of patients with oropharyngeal cancer. N Engl J Med. 2010 Jul 1;363(1):24-35. doi: 10.1056/NEJMoa0912217. Epub 2010 Jun 7. PMID 20530316
- [Background] Stanley MA. Immune responses to human papilloma viruses. Indian J Med Res. 2009 Sep;130(3):266-76. PMID 19901436
- [Background] Lehoux M, D'Abramo CM, Archambault J. Molecular mechanisms of human papillomavirus-induced carcinogenesis. Public Health Genomics. 2009;12(5-6):268-80. doi: 10.1159/000214918. Epub 2009 Aug 11. PMID 19684440
- [Background] de Vos van Steenwijk PJ, Heusinkveld M, Ramwadhdoebe TH, Lowik MJ, van der Hulst JM, Goedemans R, Piersma SJ, Kenter GG, van der Burg SH. An unexpectedly large polyclonal repertoire of HPV-specific T cells is poised for action in patients with cervical cancer. Cancer Res. 2010 Apr 1;70(7):2707-17. doi: 10.1158/0008-5472.CAN-09-4299. Epub 2010 Mar 16. PMID 20233872
- [Background] Albers A, Abe K, Hunt J, Wang J, Lopez-Albaitero A, Schaefer C, Gooding W, Whiteside TL, Ferrone S, DeLeo A, Ferris RL. Antitumor activity of human papillomavirus type 16 E7-specific T cells against virally infected squamous cell carcinoma of the head and neck. Cancer Res. 2005 Dec 1;65(23):11146-55. doi: 10.1158/0008-5472.CAN-05-0772. PMID 16322265
- [Background] Hoffmann TK, Arsov C, Schirlau K, Bas M, Friebe-Hoffmann U, Klussmann JP, Scheckenbach K, Balz V, Bier H, Whiteside TL. T cells specific for HPV16 E7 epitopes in patients with squamous cell carcinoma of the oropharynx. Int J Cancer. 2006 Apr 15;118(8):1984-91. doi: 10.1002/ijc.21565. PMID 16284959
- [Background] Tindle RW. Immune evasion in human papillomavirus-associated cervical cancer. Nat Rev Cancer. 2002 Jan;2(1):59-65. doi: 10.1038/nrc700. PMID 11902586
- [Background] Grulich AE, van Leeuwen MT, Falster MO, Vajdic CM. Incidence of cancers in people with HIV/AIDS compared with immunosuppressed transplant recipients: a meta-analysis. Lancet. 2007 Jul 7;370(9581):59-67. doi: 10.1016/S0140-6736(07)61050-2. PMID 17617273
- [Background] Chaturvedi AK, Madeleine MM, Biggar RJ, Engels EA. Risk of human papillomavirus-associated cancers among persons with AIDS. J Natl Cancer Inst. 2009 Aug 19;101(16):1120-30. doi: 10.1093/jnci/djp205. Epub 2009 Jul 31. PMID 19648510
- [Background] Frumento G, Piazza T, Di Carlo E, Ferrini S. Targeting tumor-related immunosuppression for cancer immunotherapy. Endocr Metab Immune Disord Drug Targets. 2006 Sep;6(3):233-7. doi: 10.2174/187153006778250019. PMID 17017974
- [Background] Kim R, Emi M, Tanabe K, Arihiro K. Tumor-driven evolution of immunosuppressive networks during malignant progression. Cancer Res. 2006 Jun 1;66(11):5527-36. doi: 10.1158/0008-5472.CAN-05-4128. PMID 16740684
- [Background] Marigo I, Dolcetti L, Serafini P, Zanovello P, Bronte V. Tumor-induced tolerance and immune suppression by myeloid derived suppressor cells. Immunol Rev. 2008 Apr;222:162-79. doi: 10.1111/j.1600-065X.2008.00602.x. PMID 18364001
- [Background] Gabrilovich DI, Nagaraj S. Myeloid-derived suppressor cells as regulators of the immune system. Nat Rev Immunol. 2009 Mar;9(3):162-74. doi: 10.1038/nri2506. PMID 19197294
- [Background] Almand B, Clark JI, Nikitina E, van Beynen J, English NR, Knight SC, Carbone DP, Gabrilovich DI. Increased production of immature myeloid cells in cancer patients: a mechanism of immunosuppression in cancer. J Immunol. 2001 Jan 1;166(1):678-89. doi: 10.4049/jimmunol.166.1.678. PMID 11123353
- [Background] Diaz-Montero CM, Salem ML, Nishimura MI, Garrett-Mayer E, Cole DJ, Montero AJ. Increased circulating myeloid-derived suppressor cells correlate with clinical cancer stage, metastatic tumor burden, and doxorubicin-cyclophosphamide chemotherapy. Cancer Immunol Immunother. 2009 Jan;58(1):49-59. doi: 10.1007/s00262-008-0523-4. Epub 2008 Apr 30. PMID 18446337
- [Background] Sica A, Bronte V. Altered macrophage differentiation and immune dysfunction in tumor development. J Clin Invest. 2007 May;117(5):1155-66. doi: 10.1172/JCI31422. PMID 17476345
- [Background] Haile LA, von Wasielewski R, Gamrekelashvili J, Kruger C, Bachmann O, Westendorf AM, Buer J, Liblau R, Manns MP, Korangy F, Greten TF. Myeloid-derived suppressor cells in inflammatory bowel disease: a new immunoregulatory pathway. Gastroenterology. 2008 Sep;135(3):871-81, 881.e1-5. doi: 10.1053/j.gastro.2008.06.032. Epub 2008 Jun 12. PMID 18674538
- [Background] Delano MJ, Scumpia PO, Weinstein JS, Coco D, Nagaraj S, Kelly-Scumpia KM, O'Malley KA, Wynn JL, Antonenko S, Al-Quran SZ, Swan R, Chung CS, Atkinson MA, Ramphal R, Gabrilovich DI, Reeves WH, Ayala A, Phillips J, Laface D, Heyworth PG, Clare-Salzler M, Moldawer LL. MyD88-dependent expansion of an immature GR-1(+)CD11b(+) population induces T cell suppression and Th2 polarization in sepsis. J Exp Med. 2007 Jun 11;204(6):1463-74. doi: 10.1084/jem.20062602. Epub 2007 Jun 4. PMID 17548519
- [Background] Brys L, Beschin A, Raes G, Ghassabeh GH, Noel W, Brandt J, Brombacher F, De Baetselier P. Reactive oxygen species and 12/15-lipoxygenase contribute to the antiproliferative capacity of alternatively activated myeloid cells elicited during helminth infection. J Immunol. 2005 May 15;174(10):6095-104. doi: 10.4049/jimmunol.174.10.6095. PMID 15879104
- [Background] Angulo I, de las Heras FG, Garcia-Bustos JF, Gargallo D, Munoz-Fernandez MA, Fresno M. Nitric oxide-producing CD11b(+)Ly-6G(Gr-1)(+)CD31(ER-MP12)(+) cells in the spleen of cyclophosphamide-treated mice: implications for T-cell responses in immunosuppressed mice. Blood. 2000 Jan 1;95(1):212-20. PMID 10607705
- [Background] Zhu B, Bando Y, Xiao S, Yang K, Anderson AC, Kuchroo VK, Khoury SJ. CD11b+Ly-6C(hi) suppressive monocytes in experimental autoimmune encephalomyelitis. J Immunol. 2007 Oct 15;179(8):5228-37. doi: 10.4049/jimmunol.179.8.5228. PMID 17911608
- [Background] Kerr EC, Raveney BJ, Copland DA, Dick AD, Nicholson LB. Analysis of retinal cellular infiltrate in experimental autoimmune uveoretinitis reveals multiple regulatory cell populations. J Autoimmun. 2008 Dec;31(4):354-61. doi: 10.1016/j.jaut.2008.08.006. Epub 2008 Oct 5. PMID 18838247
- [Background] Makarenkova VP, Bansal V, Matta BM, Perez LA, Ochoa JB. CD11b+/Gr-1+ myeloid suppressor cells cause T cell dysfunction after traumatic stress. J Immunol. 2006 Feb 15;176(4):2085-94. doi: 10.4049/jimmunol.176.4.2085. PMID 16455964
- [Background] Kusmartsev S, Nagaraj S, Gabrilovich DI. Tumor-associated CD8+ T cell tolerance induced by bone marrow-derived immature myeloid cells. J Immunol. 2005 Oct 1;175(7):4583-92. doi: 10.4049/jimmunol.175.7.4583. PMID 16177103
- [Background] Xu W, Liu LZ, Loizidou M, Ahmed M, Charles IG. The role of nitric oxide in cancer. Cell Res. 2002 Dec;12(5-6):311-20. doi: 10.1038/sj.cr.7290133. PMID 12528889
- [Background] Ambs S, Merriam WG, Ogunfusika MO, Bennett WP, Ishibe N, Hussain SP, Tzeng EE, Geller DA, Billiar TR, Harris CC. p53 and vascular endothelial growth factor regulate tumor growth of NOS2-expressing human carcinoma cells. Nat Med. 1998 Dec;4(12):1371-6. doi: 10.1038/3957. PMID 9846573
- [Background] Kao J, Packer S, Vu HL, Schwartz ME, Sung MW, Stock RG, Lo YC, Huang D, Chen SH, Cesaretti JA. Phase 1 study of concurrent sunitinib and image-guided radiotherapy followed by maintenance sunitinib for patients with oligometastases: acute toxicity and preliminary response. Cancer. 2009 Aug 1;115(15):3571-80. doi: 10.1002/cncr.24412. PMID 19536893
- [Background] Thomas KA. Vascular endothelial growth factor, a potent and selective angiogenic agent. J Biol Chem. 1996 Jan 12;271(2):603-6. doi: 10.1074/jbc.271.2.603. No abstract available. PMID 8557658
- [Background] Riedel F, Gotte K, Schwalb J, Wirtz H, Bergler W, Hormann K. Serum levels of vascular endothelial growth factor in patients with head and neck cancer. Eur Arch Otorhinolaryngol. 2000;257(6):332-6. doi: 10.1007/s004059900208. PMID 10993554
- [Background] Ambs S, Bennett WP, Merriam WG, Ogunfusika MO, Oser SM, Khan MA, Jones RT, Harris CC. Vascular endothelial growth factor and nitric oxide synthase expression in human lung cancer and the relation to p53. Br J Cancer. 1998 Jul;78(2):233-9. doi: 10.1038/bjc.1998.470. PMID 9683299
- [Background] Marrogi AJ, Travis WD, Welsh JA, Khan MA, Rahim H, Tazelaar H, Pairolero P, Trastek V, Jett J, Caporaso NE, Liotta LA, Harris CC. Nitric oxide synthase, cyclooxygenase 2, and vascular endothelial growth factor in the angiogenesis of non-small cell lung carcinoma. Clin Cancer Res. 2000 Dec;6(12):4739-44. PMID 11156228
- [Background] Brown LF, Berse B, Jackman RW, Tognazzi K, Manseau EJ, Senger DR, Dvorak HF. Expression of vascular permeability factor (vascular endothelial growth factor) and its receptors in adenocarcinomas of the gastrointestinal tract. Cancer Res. 1993 Oct 1;53(19):4727-35. PMID 8402650
- [Background] Nakamura Y, Yasuoka H, Tsujimoto M, Yang Q, Tsukiyama A, Imabun S, Nakahara M, Nakao K, Nakamura M, Mori I, Kakudo K. Clinicopathological significance of vascular endothelial growth factor-C in breast carcinoma with long-term follow-up. Mod Pathol. 2003 Apr;16(4):309-14. doi: 10.1097/01.MP.0000062858.98295.9F. PMID 12692195
- [Background] Mazzoni A, Bronte V, Visintin A, Spitzer JH, Apolloni E, Serafini P, Zanovello P, Segal DM. Myeloid suppressor lines inhibit T cell responses by an NO-dependent mechanism. J Immunol. 2002 Jan 15;168(2):689-95. doi: 10.4049/jimmunol.168.2.689. PMID 11777962
- [Background] Kusmartsev S, Gabrilovich DI. Immature myeloid cells and cancer-associated immune suppression. Cancer Immunol Immunother. 2002 Aug;51(6):293-8. doi: 10.1007/s00262-002-0280-8. Epub 2002 Apr 24. PMID 12111117
- [Background] Bunt SK, Yang L, Sinha P, Clements VK, Leips J, Ostrand-Rosenberg S. Reduced inflammation in the tumor microenvironment delays the accumulation of myeloid-derived suppressor cells and limits tumor progression. Cancer Res. 2007 Oct 15;67(20):10019-26. doi: 10.1158/0008-5472.CAN-07-2354. PMID 17942936
- [Background] Liu WM, Fowler DW, Smith P, Dalgleish AG. Pre-treatment with chemotherapy can enhance the antigenicity and immunogenicity of tumours by promoting adaptive immune responses. Br J Cancer. 2010 Jan 5;102(1):115-23. doi: 10.1038/sj.bjc.6605465. Epub 2009 Dec 8. PMID 19997099
- [Background] Nowak AK, Lake RA, Robinson BW. Combined chemoimmunotherapy of solid tumours: improving vaccines? Adv Drug Deliv Rev. 2006 Oct 1;58(8):975-90. doi: 10.1016/j.addr.2006.04.002. Epub 2006 Aug 15. PMID 17005292
- [Background] Vu HL, Sikora AG, Fu S, Kao J. HPV-induced oropharyngeal cancer, immune response and response to therapy. Cancer Lett. 2010 Feb 28;288(2):149-55. doi: 10.1016/j.canlet.2009.06.026. Epub 2009 Jul 22. PMID 19628331
- [Background] Smeets SJ, Hesselink AT, Speel EJ, Haesevoets A, Snijders PJ, Pawlita M, Meijer CJ, Braakhuis BJ, Leemans CR, Brakenhoff RH. A novel algorithm for reliable detection of human papillomavirus in paraffin embedded head and neck cancer specimen. Int J Cancer. 2007 Dec 1;121(11):2465-72. doi: 10.1002/ijc.22980. PMID 17680565
- [Background] Kadish AS, Ho GY, Burk RD, Wang Y, Romney SL, Ledwidge R, Angeletti RH. Lymphoproliferative responses to human papillomavirus (HPV) type 16 proteins E6 and E7: outcome of HPV infection and associated neoplasia. J Natl Cancer Inst. 1997 Sep 3;89(17):1285-93. doi: 10.1093/jnci/89.17.1285. PMID 9293919
- [Background] Kadish AS, Timmins P, Wang Y, Ho GY, Burk RD, Ketz J, He W, Romney SL, Johnson A, Angeletti R, Abadi M; Albert Einstein Cervix Dysplasia Clinical Consortium. Regression of cervical intraepithelial neoplasia and loss of human papillomavirus (HPV) infection is associated with cell-mediated immune responses to an HPV type 16 E7 peptide. Cancer Epidemiol Biomarkers Prev. 2002 May;11(5):483-8. PMID 12010863
- [Background] Santin AD, Hermonat PL, Ravaggi A, Chiriva-Internati M, Pecorelli S, Parham GP. Radiation-enhanced expression of E6/E7 transforming oncogenes of human papillomavirus-16 in human cervical carcinoma. Cancer. 1998 Dec 1;83(11):2346-52. doi: 10.1002/(sici)1097-0142(19981201)83:113.0.co;2-g. PMID 9840534
- [Background] Eric A, Juranic Z, Tisma N, Plesinac V, Borojevic N, Jovanovic D, Milovanovic Z, Gavrilovic D, Ilic B. Radiotherapy-induced changes of peripheral blood lymphocyte subpopulations in cervical cancer patients: relationship to clinical response. J BUON. 2009 Jan-Mar;14(1):79-83. PMID 19373951
- [Background] Delgado FG, Martinez E, Cespedes MA, Bravo MM, Navas MC, Combita Rojas AL. Increase of human papillomavirus-16 E7-specific T helper type 1 response in peripheral blood of cervical cancer patients after radiotherapy. Immunology. 2009 Apr;126(4):523-34. doi: 10.1111/j.1365-2567.2008.02912.x. Epub 2008 Sep 5. PMID 18778290